CLINICAL TRIAL: NCT06291948
Title: A Randomized, Double-blind, Parallel Groups, Phase 1 Clinical Study Comparing the Pharmacokinetic, Safety and Immunogenicity of Adalimumab in Healthy Subjects
Brief Title: A Clinical Study With Adalimumab Biosimilar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Richmond S.A.C.I.F. (Industry)
Collaborators: FP Clinical Pharma S.R.L. (Industry); Custom Biologics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 0225
Record Dates: First submitted 2023-12-04; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Pharmacokinetics; Safety Issues
Keywords: adalimumab; Biosimilar; Rheumatoid arthritis; Bioequivalence; Immunogenicity; Safety; Enthesitis-related arthritis; Psoriatic arthritis; Ankylosing Spondylitis (AS); Non-radiographic axial spondyloarthritis; Crohn's disease; Plaque psoriasis; Ulcerative colitis; Hidradenitis suppurativa; Behcet's Intestinal Disease; Non-infectious uveitis; Adults, healthy, of both sexes
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile; Arthritis, Psoriatic; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Crohn Disease; Colitis, Ulcerative; Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: A Randomized, Double Blind, Parallel groups, Phase 1 Clinical Study comparing the Pharmacokinetic, Safety and Immunogenicity of Adalimumab in Healthy Subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, investigators, Sponsor, monitor, analytical center, and data analyst will be unaware of assigned treatments.
  Each product in its original primary packaging will be blinded and labeled with a fantasy name "Product A" or "Product B".
  The link between "Product A or B" with the Test Product or Reference Product will be kept in two separate copies in a sealed envelope. One copy will remain with the Sponsor and the other will be provided to the Principal Investigator. The envelope may only be opened in the event of a medical emergency. The investigator must follow the trial's randomization procedures, and must ensure that the code is broken only in accordance with the protocol. The investigator must promptly document and explain to the Sponsor should the identity of the investigational product be revealed (whether accidentally or due to a serious adverse event).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humira® (adalimumab) AC Pen [Reference Product] (Active Comparator): A single subcutaneous dose of 40 mg of the Reference Product- Humira® AC Pen [Reference Product]
  Interventions: Biological: Humira® (adalimumab) AC Pen [Reference Product]
- Adalimumab Richmond [Test Product] (Active Comparator): A single subcutaneous dose of 40 mg of the Test Product- Adalimumab Richmond [Test Product]
  Interventions: Biological: Adalimumab Richmond [Test Product]

INTERVENTIONS:
Biological: Humira® (adalimumab) AC Pen [Reference Product] — A single subcutaneous dose
  Arms: Humira® (adalimumab) AC Pen [Reference Product]
Biological: Adalimumab Richmond [Test Product] — A single subcutaneous dose
  Arms: Adalimumab Richmond [Test Product]

SUMMARY:
The study aims to evaluate the pharmacokinetic profile, safety profile, and immunogenic potential of adalimumab of a new citrate-free formulation of adalimumab (Adalimumab Richmond) [Test Product] vs. Humira® AC Pen [Reference Product]

DETAILED DESCRIPTION:
This is a phase 1 pharmacokinetic, safety and immunogenicity comparative, single-dose, double-blind, randomized, balanced parallel-group clinical study conducted in healthy subjects of both sexes.

Blood samples are collected for up to 71 days to determine the quantification of adalimumab and for 12 months for antidrug antibody detection. Safety and tolerability are also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent

   * Study subjects must be able to understand and comply with the protocol.
   * Study subjects must be willing and able to provide written informed consent.
2. Target population

   * Study subjects, volunteers, adults, healthy.
   * Study subjects with normal physical examination or with findings that, in the investigator's opinion, have no clinical relevance.
   * Study subjects whose safety and complementary laboratory tests are within normal values or who, in the investigator's opinion, have no clinical relevance.
   * Body mass index between 19 and 27 kg/m2 at the screening visit.
   * Study subjects preferably non-smokers. Smokers must refrain from smoking during the clinical research protocol.
   * Study subjects should not have a history of drug and/or alcohol abuse.
3. Age and gender

   * Women and men, from 21 to 55 years of age.
   * Women must not be pregnant. Women must use adequate non-hormonal contraception to prevent pregnancy throughout the clinical investigation protocol [and for a period of not less than 5 months after the last dose of the investigational product].
   * Men with a partner of childbearing potential must agree that their partner use adequate contraception prior to study entry [and for a period of not less than 5 months after the last dose of investigational product]. An adequate contraceptive method is understood to be any hormonal contraceptive method or intrauterine device (which must be established before the start of the study) and the use of a spermicide as a barrier method. Use of a barrier method alone or sexual abstinence is not considered appropriate.
   * Subjects must agree not to donate sperm during the study and for 5 months after treatment.

Exclusion Criteria:

1. Medical history and concurrent illnesses

   * History of cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, endocrine-metabolic, neurological disease or conditions of psychiatric origin (depressive disorders, in particular) at the time of taking the history and physical examination during the first visit of the clinical research protocol.
   * History of allergic drug reactions of any kind.
   * History of orthostatic hypotension.
   * Blood donation within 3 months prior to screening.
   * Participation in another clinical pharmacology study in the last 3 months.
   * History and/or current history of clinically significant diseases or disorders that, in the investigator's opinion, may prevent the participation of the study subject for safety reasons or that may influence the results of the study as well as the capacity of the study subject. to participate in the clinical research protocol.
   * History of hypersensitivity to adalimumab and/or any of the excipients.
   * Previous exposure to a biological product.
2. Physical findings and laboratory tests

   * Cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, endocrine-metabolic, neurological disease or conditions of psychiatric origin (depressive disorders, in particular).
   * Clinically significant abnormalities in any laboratory tests
   * Positive serology for HIV, hepatitis B, hepatitis C.
3. Sex and reproductive condition

   - Women of childbearing potential who are unwilling or unable to use an adequate non-hormonal method of contraception throughout the clinical investigation protocol [and for a period of not less than 5 months after the last dose of the investigational product].
4. Allergies, adverse drug reactions and contraindications

   - Study subjects with allergies, adverse drug reactions or contraindications to therapy.
5. Prohibited treatments and/or therapies

   - The study subjects must have suspended any drug treatments at least 2 weeks before starting this clinical research protocol.
6. Other exclusion criteria

   * Non-cooperative study subjects.
   * Study subjects employed by the investigator or the Clinical Pharmacokinetic Research Unit, with direct participation in the clinical investigation protocol or other clinical protocols under the direction of the Investigator or the Clinical Pharmacokinetic Research Unit.

The eligibility criteria for this clinical research protocol have been considered to guarantee the safety of the study subjects and ensure that their results can be used.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Peak Serum Concentration of adalimumab (Cmax) | Pre-dose: 0.00; Post-dose: 4.0; 8.0; 12.0; 24.0; 48.0; 72.0; 96.0; 120.0; 144.0; 168.0; 192.0; 336.0; 504.0; 672.0; 840.0; 1008.0; 1344.0; 1680.0 hours
  Cmax will be obtained directly from the serum concentration-time curve
Area Under the Serum Concentration-time Curve of adalimumab (ABC0-t) | Day 1 to Day 71
  Area under the serum concentration-time curve from time zero to the last experimental point, will be calculated by the trapezoidal rule
Area Under the Serum Concentration- Time Curve ob adalimumab (ABC0-∞) | Day 1 to Day 71
  Area under the serum concentration- time curve from time zero to infinity

SECONDARY OUTCOMES:
Number of samples with positive Anti-adalimumab serum antibodies | Screening, post dose: 672.0 hours, 1680.0 hours, 12 months
  Anti-adalimumab serum antibodies detection

OTHER OUTCOMES:
Adverse Events | Day 1 to Day 71
  Report the nature and incidence of adverse events and the eventual suspension or abandonment of the study or the participation of a study subject.
Number of positive Anti-adalimumab serum samples with neutralizing capacity | Screening, post dose: 672.0 hours, 1680.0 hours, 12 months
  To determine the neutralizing capacity of anti-adalimumab antibody positive samples

CONTACTS AND LOCATIONS:
Overall Officials: Ethel C. Feleder, MD, Principal Investigator — FP Clinical Pharma S.R.L.
Locations (1):
- FP Clinical Pharma S.R.L., Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Background] Lembach J, Skerjanec A, Haliduola H, Hass N, von Richter O, Fuhr R, Koernicke T. Randomized, Double-Blind, Single-Dose, Three-Arm Parallel Trial to Determine the Pharmacokinetics and Safety of GP2017, EU- and US-Adalimumab in Healthy Male Subjects. Arthritis Rheumatol, 69(10), 2017
- [Background] Wynne C, Altendorfer M, Sonderegger I, Gheyle L, Ellis-Pegler R, Buschke S, Lang B, Assudani D, Athalye S, Czeloth N. Bioequivalence, safety and immunogenicity of BI 695501, an adalimumab biosimilar candidate, compared with the reference biologic in a randomized, double-blind, active comparator phase I clinical study (VOLTAIRE(R)-PK) in healthy subjects. Expert Opin Investig Drugs. 2016 Dec;25(12):1361-1370. doi: 10.1080/13543784.2016.1255724. PMID 27813422
- See also: PubMed ID: 11590294 — https://pubmed.ncbi.nlm.nih.gov/11590294/
- See also: A Randomized, Double-Blind, Single-Dose, Three-Arm Parallel Trial to Determine the Pharmacokinetics and Safety of GP2017, EU- and US-Adalimumab in Healthy Male Subjects. — https://acrabstracts.org/abstract/randomized-double-blind-single-dose-three-arm-parallel-trial-to-determine-the-pharmacokinetics-and-safety-of-gp2017-eu-and-us-adalimumab-in-healthy-male-subjects/
- See also: PubMed ID: 27813422 — https://pubmed.ncbi.nlm.nih.gov/27813422/